CLINICAL TRIAL: NCT02933905
Title: Influence of the Vitreomacular Interface on the Progression of the Diabetic Macular Edema After Anti-VEGF Injection
Status: Completed | Type: Observational
Sponsor: Fundació Institut Germans Trias i Pujol (Other)
Responsible Party: Principal Investigator, Xavier Valldeperas, MD, PhD, FEBO, Fundació Institut Germans Trias i Pujol
Other Study IDs: OFT-RAN-2013-01
Record Dates: First submitted 2016-10-12; First posted 2016-10-14 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Diabetic Macular Edema; Vitreomacular Interface; Anti-VEGF Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Non-PVD subjects: Patients with no PVD on SD-OCT at basal visit
  Interventions: Drug: Intravitreal Ranibizumab injection
- PVD subjects: Patients with PVD on SD-OCT at basal visit
  Interventions: Drug: Intravitreal Ranibizumab injection

INTERVENTIONS:
Drug: Intravitreal Ranibizumab injection

SUMMARY:
Influence of the vitreomacular interface on the progression of diabetic macular edema after treatment with intravitreal injection of vascular endothelial growth factor inhibitors

ELIGIBILITY:
Inclusion Criteria:

* diabetic macular edema treatable with antiangiogenic drugs

Exclusion Criteria:

* age under 18
* cardiovascular events during the last year
* previous vitrectomy
* previous macular edema treatment during the last 4 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetic macular edema
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in best-corrected visual acuity | One year

SECONDARY OUTCOMES:
Change in central macular thickness | One year
Number of ranibizumab injections | One year